CLINICAL TRIAL: NCT05831371
Title: Discard the Curative Causes of Late Onset Epilepsy: the Role of Brain 18F-FDG PET
Acronym: EPITEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, TYVAERT Louise, Pr, Central Hospital, Nancy, France
Other Study IDs: 2023PI065
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Late Onset Epilepsy; Alzheimer Disease
Keywords: FDG PET; cognitive prognosis
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TEP FDG — FDG TEP peformed in clinical routine

SUMMARY:
Etiology and cognitive prognosis in late onset epilepsy differ from young adults epilepsy. At the epilepsy onset, this is crucial to detect potential curative/treatable brain disorders. After classical investigation including morphological brain imaging, EEG, clinical assessment, which added value may have brain FDG PET in the diagnosis and prognosis evaluation?

ELIGIBILITY:
Inclusion Criteria:

* late onset épilepsy patients without lesion
* epilepsy followed at the CHRU Nancy france

Exclusion Criteria:

* epilepsy explained by cortical lesion
* severe psychiatric disorders
* severe addiction (alcool, drugs)
* no FDG TEP performed
* no neuropsychological assessement after 2 years epilepsy onset

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non lesional late onset epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2023-05-02 (Estimated); Primary Completion 2023-08-02 (Estimated); Study Completion 2023-09-02 (Estimated)

PRIMARY OUTCOMES:
diagnostic performances | 2 years after epilepsy onset
  sensibility, specificty, accurracy

SECONDARY OUTCOMES:
cognitive prognosis performances | 2 years after epilepsy onset
  sensibility, specificty, accurracy

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No